CLINICAL TRIAL: NCT06038071
Title: Efficacy and Safety of Family Mid-upper Arm Circumference (MUAC) After Recovery From Severe and Moderate Acute Malnutrition
Brief Title: Family Mid-Upper Arm Circumference (MUAC) Follow-up After Recovery From Acute Malnutrition (MODAM-fMUAC)
Acronym: MODAM-fMUAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Action Against Hunger USA (Other)
Collaborators: University of Washington (Other); Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Heather Stobaugh, Senior Research and Learning Specialist, Action Against Hunger USA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MODAM-fMUAC
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Severe Acute Malnutrition; Moderate Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): nutrition, IYCF, and WASH education at discharge, followed by regular community-based screenings led by health extension workers, with one final visit scheduled at 6 months after discharge
  Interventions: Other: nutrition, IYCF, WASH education
- scheduled followup (Active Comparator): standard of care plus scheduled follow-up visits at 1 month, 3 months, 6 months after discharge
  Interventions: Other: nutrition, IYCF, WASH education; Other: scheduled anthropometric screening
- family MUAC (Experimental): standard of care plus Family MUAC training for the primary caregiver present at the time of recovery, with one final visit scheduled at 6 months after discharge
  Interventions: Other: nutrition, IYCF, WASH education; Other: family MUAC

INTERVENTIONS:
Other: nutrition, IYCF, WASH education — nutrition, IYCF, WASH education
Other: scheduled anthropometric screening — anthropometric screening by health care workers at 1, 3, and 6 months
  Arms: scheduled followup
Other: family MUAC — family MUAC training for the primary caregiver present at the time of recovery
  Arms: family MUAC

SUMMARY:
Protocols for the community-based management of acute malnutrition (CMAM) have not changed significantly for more than 20 years, with relatively complex treatment protocols and persistent supply chain challenges that have limited overall program coverage, leaving millions of malnourished children without care annually. The overarching goal of this research project is to simultaneously test two novel simplified approaches in CMAM with potential to improve program coverage. The simplified approach includes two parallel clinical trials for SAM and MAM treatment. For the Family MUAC follow-up study, children who recover from these two parallel clinical trials will be enrolled in trial to test the effectiveness of MUAC screening at home by the child's caregivers as a self-referral strategy, compared to a scheduled health facility-led strategy and the standard of care of community-based follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* children 6-59 months of old who recovered from SAM or MAM following treatment in either the MODAM-SAM or MODAM-MAM trials

Exclusion Criteria:

* caregiver not planning on remaining in the local area for the subsequent 6 months

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3600 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
number of episodes of relapse to acute malnutrition identified | 6 months

SECONDARY OUTCOMES:
weight-for-height Z-score (WHZ) at time relapse to acute malnutrition identified | 6 months
mid-upper arm circumference (MUAC) at time relapse to acute malnutrition identified | 6 months
number of episodes of relapse to edematous malnutrition / kwashiorkor identified | 6 months
recovery rates following treatment of relapse to acute malnutrition | 6 months
mortality | 6 months
hospitalization | 6 months
loss to follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heather C Stobaugh, Principal Investigator — Action Against Hunger USA; Indi Trehan, MD MPH DTM&H, Principal Investigator — University of Washington; Yosef B Asefaw, MSc, Principal Investigator — Ethiopian Public Health Institute
Locations (3):
- Ethiopia (3):
  - Sekota, Sekota, Amhara
  - Teltele, Teltelē, Oromiya
  - Gode, Gode, Somali

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Trehan I, Beyene Y, Darsene H, Adams BS, Wrabel M, Gizaw G, Legese LA, Cichon B, Chitekwe S, Shellemew MW, Tessema M, Stobaugh HC. The Modified Dosages for Acute Malnutrition (MODAM) study: protocol for three integrated randomized controlled trials of novel approaches for the management of childhood wasting in Ethiopia. BMC Nutr. 2025 Apr 8;11(1):71. doi: 10.1186/s40795-025-01054-w. PMID 40200326